CLINICAL TRIAL: NCT00616057
Title: Evaluation of Fructans Supplementation on Parameters of Metabolic Syndrome
Acronym: FRUCTOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007/21/NOV/300; B40320072930
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Obesity
Keywords: fructans supplementation
MeSH Terms: conditions — Obesity | interventions — Inulin; oligofructose; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Placebo Comparator): Maltodextrin, non digestible carbohydrate
  Interventions: Dietary Supplement: maltodextrin
- A (Experimental): fructans, non digestible carbohydrates fermented in the caeco-colon
  Interventions: Dietary Supplement: Synergy 1

INTERVENTIONS:
Dietary Supplement: Synergy 1 — 8 grams/day during the first week and then 8 grams twice a day during 3 months
  Other Names: inulin; oligofructose
  Arms: A
Dietary Supplement: maltodextrin — 8 grams/day during the first week and then 8 grams twice a day during 3 months
  Arms: B

SUMMARY:
Obesity is constantly increasing, causing an important risk to develop diseases such as heart disease, diabetes,... Some recent studies have shown that obese people present modifications of colon microflora and a low-grade inflammation.

In our laboratory, we have demonstrated that the intake of fructans lessens dietary intake, body weight gain, adipose tissue accumulation and steatosis in rodents. These effects lead to an improvement of insulin resistance and hyperglycemia in diabetic rats and mice. Fructans are also able to restore the microflora disturbed by a high fat diet and to prevent endotoxemia. Moreover, studies have shown that fructans intake promotes satiety (Cani et al, Diabetes 2007) and or decreases fat mass (Abrams et al, Journal of Pediatrics 2007) in healthy human. An intervention study in obese patients is thus needed to study the effects of fructans in the target population.

ELIGIBILITY:
Inclusion Criteria:

* BMI>30 kg/m2

Exclusion Criteria:

* acute or chronic evoluting disease
* alcohol consumption > 30 units/week
* more than 30 minutes of sports 3 times/week
* usual consumption of pre/probiotics or fibers supplement
* recent consumption of antibiotics
* slimming diet or unusual diet
* pregnant women
* anti-diabetics drugs ou slimming drugs
* previous bariatric surgery
* severe oesophagus reflux

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-02; Primary Completion 2010-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
gut microbiota composition | 3 months
  HITChip analysis (phylogenetic profiling by DNA microarray)

SECONDARY OUTCOMES:
gut microbial-related metabolites (in urine and plasma) | 3 months
  NMR spectroscopic analysis of urine and plasma metabolic profiles
metabolic parameters (weight, BMI, glycemia, fat mass,...) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Thissen Jean-Paul, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint Luc, Brussels, Branbant Wallon, Belgium

REFERENCES:
- [Derived] Salazar N, Dewulf EM, Neyrinck AM, Bindels LB, Cani PD, Mahillon J, de Vos WM, Thissen JP, Gueimonde M, de Los Reyes-Gavilan CG, Delzenne NM. Inulin-type fructans modulate intestinal Bifidobacterium species populations and decrease fecal short-chain fatty acids in obese women. Clin Nutr. 2015 Jun;34(3):501-7. doi: 10.1016/j.clnu.2014.06.001. Epub 2014 Jun 11. PMID 24969566